CLINICAL TRIAL: NCT03388788
Title: Circadian Mechanisms of Cardiovascular Risk in Obesity
Brief Title: Body Weight, Sleep, and Heart Health
Status: Active, not recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Steven A. Shea, Director, Oregon Health and Science University
Other Study IDs: IRB00017489; R01HL140577 (NIH); KL2TR002370 (NIH)
Record Dates: First submitted 2017-12-20; First posted 2018-01-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Risk Factor; Circadian Dysregulation; Obesity
MeSH Terms: conditions — Chronobiology Disorders; Obesity | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Weight: Healthy lean controls [18.5<BMI<25 kg/m2 and waist circumference <94/80 cm (men/women respectively)] will participate in a 5-day circadian study protocol with numerous repeated cardiovascular measures across the circadian cycle. Drugs are used as part of physiological monitoring and not as interventions including imaging using radiopharmaceuticals (11C-meta-hydroxyephedrine, and 11C-CGP12177).
  Interventions: Combination Product: Positron Emission Tomography (PET) scanning of cardiac function at 3 time points across the 24 hour circadian cycle
- Overweight: Healthy obese [30≤BMI<40 and waist circumference ≥94/80 (men and women respectively)] Healthy lean controls [18.5<BMI<25 kg/m2 and waist circumference <94/80 cm (men/women respectively)] will participate in a 5-day circadian study protocol with numerous repeated cardiovascular measures across the circadian cycle. Drugs are used as part of physiological monitoring and not as interventions including imaging using radiopharmaceuticals (11C-meta-hydroxyephedrine, and 11C-CGP12177).
  Interventions: Combination Product: Positron Emission Tomography (PET) scanning of cardiac function at 3 time points across the 24 hour circadian cycle

INTERVENTIONS:
Combination Product: Positron Emission Tomography (PET) scanning of cardiac function at 3 time points across the 24 hour circadian cycle — Drugs are used for as part of physiological monitoring and not as interventions, including imaging using radiopharmaceuticals (11C-meta-hydroxyephedrine, and 11C-CGP12177).
  Other Names: PET scanning

SUMMARY:
A multidisciplinary investigation examining the circadian mechanisms regulating cardiovascular (CV) risk, with an additional focus on obesity. Specifically, in a valid circadian protocol, the investigators aim to study resting cardiovascular risk markers and the reactivity of circadian rhythms in these risk markers to standardized stressors. It is intended to compare results in lean and obese individuals to determine if there are specific risks across the circadian cycle specific to obesity. Furthermore, using an exploratory approach, the investigators propose to explore impairment in pre/post synaptic function in the cardiac left ventricle.

DETAILED DESCRIPTION:
Overall, these studies will help us answer whether the circadian system predispose individuals to increased CV disease risk - particularly around the vulnerable morning period, and whether these risks differ with obesity. The results will serve as a foundation for clinical trials of appropriately timed dosing of medications targeting aspects of the CV system that increase effectiveness while decreasing side effects, and may have particular relevance to management of CV risk in people with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Ages 25-65
* Lean and overweight (BMI 18.5-40kg/m2)
* Habitually sedentary

Exclusion Criteria:

* History of smoking/tobacco use
* Insomnia
* Moderate to severe obstructive sleep apnea.
* Prior shift work within 6 months prior to the study.
* Prescription medications
* Drugs of abuse
* Acute, chronic, or debilitating medical condition (including diabetes, hypertension, and metabolic syndrome)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | 5 Days
  Beat-by-beat and ambulatory blood pressure measurements.

SECONDARY OUTCOMES:
Coronary Microvascular Blood Flux | 3 days
  Coronary microvascular function, measured as coronary microvascular blood flux using myocardial contrast echocardiography.
Flow Mediated Dilation (FMD) | 5 days
  FMD to measure endothelial function.
Heart Rate | 5 Days
  Heart rate via 2-channel echocardiogram (ECG)
Epinephrine | 5 days
  Venous Epinephrine to estimate sympathetic output
Norepinephrine | 5 days
  Venous Norepinephrine to estimate sympathetic output
Cortisol | 5 days
  Saliva cortisol to estimate sympathetic output

OTHER OUTCOMES:
Beta-adrenergic receptor density (Exploratory outcome) | 5 days.
  Radiolabeled agonist (11C-CGP12177) to measure beta-adrenergic receptors during PET Imaging.
Norepinephrine reuptake transport (Exploratory outcome) | 5 days.
  Radiolabeled meta-hydroxyephedrine (11C-mHED) to measure norepinephrine reuptake during PET Imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Shea, PhD, Principal Investigator — Oregon Institute of Occupational Health Sciences; Jeanne M Link, PhD, Principal Investigator — OHSU Center for Radiochemistry Research
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT03388788/Prot_SAP_000.pdf